CLINICAL TRIAL: NCT04314206
Title: A Randomized, Double-Blind, Placebo-Controlled, Sequential Group, Dose-Escalation Study to Evaluate the Safety and Pharmacokinetics of Single and Repeat Doses of VNRX-5024 Administered Orally for 10 Days in Healthy Adult Volunteers
Brief Title: VNRX-5024 Safety and PK in Healthy Adult Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Basilea Pharmaceutica (Industry)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Basic Science
Other Study IDs: VNRX-5024-101; 272201600029C-P00007-9999-2 (NIH); 17-0004 (Other: DMID)
Record Dates: First submitted 2020-03-16; First posted 2020-03-19 (Actual); Last update posted 2025-12-03 (Actual); Status verified 2025-11

CONDITIONS: Healthy Subjects

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- VNRX-5024 (Experimental): Capsule formulation
  Interventions: Drug: VNRX-5024
- Placebo (Placebo Comparator): Placebo for VNRX-5024
  Interventions: Drug: Placebo for VNRX-5024

INTERVENTIONS:
Drug: VNRX-5024 — Part 1: one dose
  Part 2:
  Cohort 1: 10 doses (once a day for 10 days) Cohort 2: 19 doses (once every 12 hours [q12h] dosing for 9 days with a single morning dose on Day 10) Cohort 3: 28 doses (once every 8 hours [q8h] dosing for 9 days with a single morning dose on Day 10)
  Arms: VNRX-5024
Drug: Placebo for VNRX-5024 — Part 1: one dose
  Part 2:
  Cohort 1: 10 doses (once a day for 10 days) Cohort 2: 19 doses (once every 12 hours [q12h] dosing for 9 days with a single morning dose on Day 10) Cohort 3: 28 doses (once every 8 hours [q8h] dosing for 9 days with a single morning dose on Day 10)
  Arms: Placebo

SUMMARY:
This is a 2-part dose-ranging study to evaluate the safety and pharmacokinetics of escalating doses of VNRX-5024. Subjects will be enrolled in one of three dose cohorts. They will receive a single dose on Day 1 in Part 1 and will proceed into the multiple dose Part 2 of the study after safety assessments and PK samples are collected. In the multiple dose part of the study, subjects will receive multiple doses of VNRX-5024 for 10 days.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy adults 18-55 years
2. Males or non-pregnant, non-lactating females
3. Body mass index (BMI): ≥18.5 kg/m2 and ≤32.0 kg/m2
4. Normal blood pressure
5. Normal lab tests

Exclusion Criteria:

1. Current cardiovascular, respiratory, hepatic, renal, gastrointestinal, endocrine, autoimmune, hematologic, neoplastic, or neurological disorder
2. History of drug allergy or hypersensitivity to penicillin, cephalosporin, or beta-lactam antibacterial drug
3. Use of antacid medications
4. Abnormal ECG or history of clinically significant abnormal rhythm disorder
5. Positive alcohol, drug, or tobacco use/test

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2020-07-27 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
Number of subjects with adverse events | Day 19

SECONDARY OUTCOMES:
Part 1: AUC0-tau | Days 1-2
Part 2: AUC0-tau | Days 3-12
Part 1: Cmax | Days 1-2
Part 2: Cmax | Days 3-12
Part 1: tmax | Days 1-2
Part 2: tmax | Days 3-12
Part 1: CLr | Days 1-2
Part 2: CLr | Days 3-12

CONTACTS AND LOCATIONS:
Overall Officials: Kamal Hamed, MD, Study Director — Basilea Pharmaceutica International Ltd, Allschwil
Locations (1):
- PRA Health Sciences - Early Development Services, Groningen, Netherlands

REFERENCES:
- [Derived] Dorr MB, de Oliveira CF, van de Wetering J, Lowe K, Sabato P, Winchell G, Chen H, McGovern PC. Pharmacokinetics and safety of single and repeat doses of ceftibuten in healthy participants: a phase 1 dose escalation study. Antimicrob Agents Chemother. 2025 Sep 3;69(9):e0008725. doi: 10.1128/aac.00087-25. Epub 2025 Aug 5. PMID 40762485